CLINICAL TRIAL: NCT00075426
Title: A Pilot Phase II Protocol Of Arsenic Trioxide (Trisenox) In Subjects With Advanced Non-Small Cell Carcinoma Of The Lung
Brief Title: Arsenic Trioxide in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 02-402; CDR0000346366
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well arsenic trioxide works in treating patients with locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and activity of arsenic trioxide in patients with locally advanced or metastatic non-small cell lung cancer.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.

Secondary

* Determine the response, in terms of objective tumor response and response duration, in patients treated with this drug.
* Determine the patterns of failure and survival in patients treated with this drug.

OUTLINE: This is a pilot study.

Patients receive arsenic trioxide IV over 1-2 hours on days 1-5 of week 1 and on days 1 and 5 of weeks 2-8 (course 1 only). Beginning with course 2 and for all subsequent courses, patients receive arsenic trioxide on days 1 and 5 of weeks 1-8. Treatment repeats every 8 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 1 additional course of therapy beyond CR. Patients achieving CR due to local consolidative therapy (surgery or radiotherapy) receive 2 additional courses of therapy beyond CR.

Patients are followed for 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 9-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC), meeting criteria for 1 of the following:

  * Locally advanced disease not amenable to radiotherapy or surgery
  * Metastatic disease
* Received at least 1 course of platinum-based (e.g., cisplatin or carboplatin) chemotherapy
* No uncontrolled central nervous system (CNS) metastases
* Ineligible for higher priority treatment protocols

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1 OR
* Zubrod Scale 0-1 OR
* South West Oncology Group (SWOG) 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* Serum glutamate oxaloacetate transaminase (SGOT) and Serum glutamate pyruvate transaminase (SGPT) no greater than 3 times normal

Renal

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 12 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No uncontrolled, clinically significant dysrhythmia
* Cardiac ejection fraction greater than 50%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Electrolytes (including magnesium) normal
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior or ongoing peripheral neuropathy grade 2 or greater
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent cytokine therapy

Chemotherapy

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens for NSCLC
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* No concurrent radiotherapy

  * Concurrent palliative or emergent radiotherapy allowed

Surgery

* More than 2 weeks since prior surgery

Other

* At least 4 weeks since prior antineoplastic agents for non-malignant conditions (e.g., methotrexate for rheumatoid arthritis)
* No concurrent antineoplastic agents for non-malignant conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennie V. Jones, MD, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States